CLINICAL TRIAL: NCT05964062
Title: Personalized Brain Functional Sectors (pBFS) Guided High-dose rTMS Therapy for Treatment-resistant Obsessive-Compulsive Disorder: A Randomized, Double-Blind, Sham-controlled Trial
Brief Title: pBFS Guided High-dose rTMS Therapy for Treatment-Resistant Obsessive-Compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLOCDpreSMA
Record Dates: First submitted 2023-07-11; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Obsessive-Compulsive Disorder; OCD
Keywords: Obsessive-Compulsive Disorder; Treatment-resistant OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active rTMS treatment (Experimental): 10 sessions of active rTMS would be delivered to the right preSMA daily, with a session of 1800 pulse.
  Interventions: Device: active rTMS treatment
- sham rTMS treatment (Sham Comparator): 5 sessions of sham rTMS would be delivered to the right preSMA daily, with a session of 1800 pulse.
  Interventions: Device: sham rTMS treatment

INTERVENTIONS:
Device: active rTMS treatment — Participants will receive 10 sessions per day of 1800 pulses per session, lasting for 5 days. Individualized targets will be generated using the pBFS method.
  Arms: active rTMS treatment
Device: sham rTMS treatment — The parameters in the sham arms are the same as the active stimulation groups. Stimulation was delivered by the same device as the active group fitted with a sham coil.
  Arms: sham rTMS treatment

SUMMARY:
The research aims to evaluate the safety and efficacy of pBFS-guided High-dose rTMS therapy targeting preSMA for patients with treatment-resistant Obsessive-Compulsive Disorder.

DETAILED DESCRIPTION:
In 2018, rTMS received approval from the U.S. Food and Drug Administration (FDA) for the treatment of OCD. Based on a systematic meta-analysis of randomized clinical trials, researchers compared the efficacy of different intervention targets (DMPFC, DLPFC, OFC, SMA) and found that targeting the anterior part of the right SMA in patients yielded the best response rates for individuals with obsessive-compulsive disorder (OCD) while targeting the DLPFC showed poor efficacy. However, the preSMA is a large region, and different nodes within this region have distinct functional connections with other areas. Thus, precise localization of neural circuitry implicated in OCD symptomatology is essential for achieving effective therapeutic interventions. Leveraging an innovative technique pBFS, the current study aims to identify individual-specific preSMA targets with functional connectivity to the attention network, enabling a more personalized and targeted approach to diagnosis and treatment for OCD patients. A novel high-dose treatment modality known as SAINT received approval from the U.S. FDA in September 2022 for managing the treatment-resistant major depressive disorder. Building upon these findings, this study hypothesizes that high-dose iTBS targeting the preSMA guided by pBFS will have a significant therapeutic effect on clinical symptoms in treatment-resistant OCD patients.

After being informed about the study and potential risks. All patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner in a 2:1 ratio to the active rTMS group, or sham-control group. Then all participants will undergo a 5-day rTMS modulation and a 1-month, 2-month 3-month follow-up visit. Patients will have a stable treatment regimen during the 5-day treatment and one-month post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized/outpatient patients aged 18-65 years (inclusive), male or female.
* Meet the diagnostic criteria of DSM-5(Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) for obsessive-compulsive disorder, and currently experiencing a first or recurrence episode.
* Total Y-BOCS score ≥20 and total HAMD score <17 before randomization.
* Before randomization, patients must have received a minimum of 2 months of maintenance treatment with SSRI medication prior to randomization, or have undergone maintenance CBT treatment with inadequate response to SSRI medication (less than 50% symptom improvement), or have previously shown inadequate response (less than 50% symptom improvement) to at least one trial of SSRI medication or cognitive-behavioral therapy. Patients currently taking medication should have been on a stable dose for 8 weeks.
* Voluntarily participate in the trial and sign informed consent. Able to comply with the planned visit, examination and treatment plan, and other study procedures.

Exclusion Criteria:

* Does not meet the inclusion criteria
* Exhibiting hoarding disorder.
* Meet DSM-5 diagnostic criteria for other mental disorders (such as schizophrenia, schizoaffective disorder, post-traumatic stress disorder, bipolar disorder, and secondary depression, etc.);
* Patients with a cardiac pacemaker, cochlear implant, or other metal foreign body and any electronic equipment implanted in the body, patients with claustrophobia and other contraindications to magnetic resonance scanning, and patients with contraindications to rTMS treatment;
* History of epilepsy (presence of at least 2 uninduced seizures more than 24 hours apart, or diagnosis of the epileptic syndrome, or seizures within the past 12 months); Or currently received medications or other treatments that will lower the seizure threshold;
* History of ECT, rTMS, light therapy within 3 months;
* Patients with organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumor, etc.) and a history of severe brain trauma as judged by the researcher;
* Patients with serious or unstable diseases of the cardiovascular, liver, kidney, blood, endocrine, neurological system, and other systems or organs.
* Female of childbearing potential who plans to become pregnant during the trial. Female that is pregnant or breastfeeding.
* Substance abuse or dependence (including alcohol misuse and drugs) within the past 6 months.
* First-degree relatives have bipolar affective disorder and schizophrenia.
* There is a significant risk of suicide (MADRS item 3 ≥ 3).
* Difficulty or inability to engage in normal communication, understand or follow instructions, and cooperate with treatment and evaluators.
* Patients currently in any clinical trials of other drugs or physical therapy ( DBS, ECT, rTMS).
* Investigators think that was inappropriate to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
response rates estimated using Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Baseline, Day 5, one-month post-treatment
  The Y-BOCS is a validated instrument stratifying the severity of obsessive episodes. This validated questionnaire was used to assess the response rate and remission rate of obsessive episodes. This research compared the response rates of Y-BOCS between groups using non-parametric rank-sum tests to assess improvement immediately post-intervention. Response is defined as a symptom improvement ≥35% on these scales;

SECONDARY OUTCOMES:
remission rate estimated using Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Baseline, Day 5, one-month post-treatment, two-month post-treatment, three-month post-treatment
  Remission was defined as a score <8.
partial response rates estimated using Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Baseline, Day 5, one-month post-treatment,two-month post-treatment, three-month post-treatment
  Partial response is defined as a symptom 35% ≥ improvement ≥25% on Y-BOCS;
cognitive change in Stroop | Baseline, Day 5
  The Stroop test can be used to measure a person's selective attention capacity and skills, processing speed, and alongside other tests to evaluate overall executive processing abilities.
cognitive change in Hopkins verbal learning test(immediate recall) | Baseline, Day 5
  The Hopkins Verbal Learning Test (HVLT-R) is one such assessment that consists of memorization of a list of words to test the ability to recall immediately after memorization
cognitive change in Trail-Making Test | Baseline, Day 5
  The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory